CLINICAL TRIAL: NCT01844544
Title: Identification and Characterization of Drug Related Problems Among Patients With Femoral Neck Fractures in an Orthopedic Ward
Brief Title: Drug Related Problems Among Patients With Femoral Neck Fractures in an Orthopedic Ward
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC130061-13CTIL
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Femoral Neck Fractures
Keywords: drug related problems; clinical pharmacist; femoral neck fractures; orthopedic patients
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients after femur neck fracture
  Interventions: Other: inspection of medical records

INTERVENTIONS:
Other: inspection of medical records

SUMMARY:
the purpose of the study is to:

1. Identify and characterize drug related problems in patients after a femur neck fracture that are hospitalized in the orthopedic department at "Meir" medical center.
2. Evaluate the contribution of a clinical pharmacist in identifying,characterizing and preventing drug related problems in patients after a femur neck fracture that are hospitalized in the orthopedic department at "Meir" medical center.

ELIGIBILITY:
Inclusion Criteria:

* patients over 64
* patients after a femoral neck fracture
* patients hospitalized in the orthopedic ward at "Meir" medical center
* patients who speak Hebrew, Russian or English

Exclusion Criteria:

* patients under 64
* patients without a femoral neck fracture
* patients who don't speak Hebrew, Russian or English

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 65 after a femoral neck fracture that are hospitalized in the orthopedic department at "Meir" medical center
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the overall number of drug related problems in patients with a femur neck fracture in the orthopedic department | participants will be followed for the duration of hospital stay, an expected average of 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel